CLINICAL TRIAL: NCT05452824
Title: Participating in Tai Chi to Reduce Anxiety and Keep up Physical Function: Implementing a Prehabilitation Intervention for Radical Prostatectomy
Brief Title: Participating in Tai Chi to Reduce Anxiety and Keep up Physical Function
Acronym: PEAK-RP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Lin Yang, Research Scientist, AHS Cancer Control Alberta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 200345
Record Dates: First submitted 2022-06-27; First posted 2022-07-11 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Single-centered, single-blind, parallel design randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Although it is not possible to blind participants or interventionists to group allocation, the random allocation sequence will be blinded from study staff conducting data management and analyses. The randomization schedule, generated by the project data analyst, will be kept by project staff who will deliver it, in a sealed envelope, to a research assistant who will then assign qualified individuals to intervention groups. Randomization will occur after informed consent is obtained and baseline assessments have been completed. Participants will be notified of their allocation through phone calls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai Chi Prehabilitation (Experimental): 8 weeks Tai Chi prehabilitation prior to radical prostatectomy
  Interventions: Other: Tai Chi Prehabilitation
- Usual Care (Placebo Comparator): Usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Tai Chi Prehabilitation — The intervention arm will be oriented to a WaQi (youthful vitality) program 8 weeks prior to their scheduled surgery date. The WaQi program uses a Tai Chi curriculum previously successfully implemented in older adults, and at the Memorial Sloan Kettering Cancer Center (MSKCC). It has an online teaching module and is uniquely suited for our study population. The program requires no difficult movement transitions, but still contains all essential parts including meditation. The WaQi program has less psychological stress and physical challenge than other exercise activities because it can be performed either sitting or standing. Intervention participants will also receive printed materials from Prostate Cancer Canada about prostate cancer management. These materials include information about how to cope with prostate cancer including pelvic floor exercise, physical activity, healthy eating, and mental wellbeing.
  Arms: Tai Chi Prehabilitation
Other: Usual care — Control arm participants will receive printed materials identical to intervention arm participants with general information on a healthy lifestyle. The control arm will receive an 8-week online Tai Chi teaching module subscription at the end of the study.
  Arms: Usual Care

SUMMARY:
The goal of the proposed project is to test the implementation strategy, in terms of feasibility and utility, of an online Tai Chi intervention as a prehabilitation model to prepare prostate cancer patients and their caregivers for radical prostatectomy (RP). The investigators' hypothesis is that, by using an online teaching module, the proposed prehabilitation model is feasible on the prostate cancer care pathway in a simple, efficient, and minimally disruptive manner. In addition, participating in the Tai Chi intervention will improve patient anxiety leading up to the RP and improve physical function as well as post-operative side-effects associated with RP.

Our primary objective is to test the feasibility of the implementation strategy from multi-stakeholder perspectives. The investigators will use mixed-methods to assess the barriers and facilitators related to implementing the online Tai Chi intervention from multi-stakeholder perspectives guided by the Consolidated Framework for Implementation Research.

Our secondary objective is to examine the effect of the Tai Chi intervention on patient outcomes at peri-RP and post-RP. The investigators will quantitatively test the effect of the intervention to reduce peri- and post-RP anxiety and improve peri- and post-RP physical function and general disease specific patient-reported outcomes.

An exploratory objective is to explore the effect of the Tai Chi intervention on surgical outcomes. The study team will quantitatively describe the difference in post-RP surgical outcomes between the intervention and control groups.

DETAILED DESCRIPTION:
The goal of the proposed project is to test the implementation strategy, in terms of feasibility and utility, of an online Tai Chi intervention as a prehabilitation model to prepare prostate cancer patients and their caregivers for radical prostatectomy (RP).

The investigators primary objective is to test the feasibility of the implementation strategy from multi-stakeholder perspectives. The study team will use mixed-methods to assess the barriers and facilitators related to implementing the online Tai Chi intervention from multi-stakeholder perspectives guided by the Consolidated Framework for Implementation Research.

The investigators secondary objective is to examine the effect of the Tai Chi intervention on patient-reported outcomes at peri-RP and post-RP. The study team will quantitatively test the effect of the intervention to reduce peri- and post-RP anxiety and improve peri- and post-RP physical function and general disease specific patient-reported outcomes.

The tertiary objective is to explore the effect of the Tai Chi intervention on surgical outcomes. We will quantitatively test the effect of the intervention in improving post-RP surgical outcomes.

Study Design and Methods:

The study team will conduct a single-centered, single-blind, parallel design, randomized controlled trial with 40 participants randomly allocated to one of two arms: usual care or 8 weeks Tai Chi prior to RP with optional caregiver participation.

The study will use a staggered participant recruitment process, in which eligible participants will undergo initial screening, consent, and baseline assessments, and then be randomized based on a 1:1 ratio allocation schedule.

The study team will recruit 30 RP patients into each of the intervention and control arms of the study. The enrollment of a caregiver of the patient is optional.

Inclusion/exclusion criteria: All participants must speak English. RP patient participants include those: (1) scheduled and awaiting RP for prostate cancer; (2) not previously treated for prostate cancer, including radiation therapy to the pelvis, major pelvic surgery, or placement of a penile implant or artificial urinary sphincter; (3) with no known urethral stricture or colostomy or chronic urinary catheterization; (4) with no medical or current psychiatric disorders that preclude their participation in the intervention; (5) with permission to exercise from their primary physicians; and (6) not currently practicing Tai Chi or related activities that involve mindfulness practice. As an option, any support person identified by the patient as a primary caregiver who is >18 years of age will be eligible. Finally, for qualitative assessment of the implementation, providers and support staff, and any individual who provides care/information for RP patients on a routine basis in a clinical setting will be eligible.

Potentially eligible patients who meet the initial inclusion criteria and individuals who are identified as the primary caregiver will be asked to participate in the study. Potential participants will be scheduled for a 1-hour virtual orientation meeting via password-protected Zoom and consent forms will be delivered to potential participants (patients and caregivers) via emails to obtain their electronic signature. At this meeting, the consent form, intervention activities and the participant responsibilities involved with the study will be discussed in depth. Participants who are clear about the study procedure and provide informed consent will be scheduled for a 1-hour in-office visit at the Prostate Cancer Center (PCC) for baseline evaluation. Prior to the in-office visit, COVID-19 screening will be performed, and symptomatic participants will be rescheduled.

Three days before participants come to the PCC, a Baseline Health Questionnaire (sociodemographic characteristics, lifestyle and gender role) and five questionnaires assessing study outcomes will be administered electronically for them to complete (Pittsburgh Sleep Quality Inventory, SF-36, Hospital Anxiety and Depression Scale, Brief Pain Inventory, the urinary and sexual domains of the Expanded Prostate Cancer Index Composite-50 [spousal version for spousal caregivers]. In addition, baseline frailty will be measured among patient participants through a modified frailty index using data extracted from electronic medical charts. One day prior to the visit, a COVID-19 screening questionnaire will be completed by telephone and if the participant is symptomatic, they will be rescheduled.

During the baseline evaluation at the PCC, hand hygiene, continuous masking and maintenance of physical distancing will be followed whenever possible. Data collection will include physical assessments of handgrip strength test and six minute walk test; and four functional tests in accordance with the US CDC STEADI program (30-second chair stand test, 4-stage balance test, timed up and go test, and orthostatic blood pressure) and instruction on how to wear an activity tracking device (Actigraph wGT3X-BT®) around their wrist for 7 days to measure usual physical activity levels. Participants will complete two self-administered questionnaires: Global Physical Activity Questionnaire assessing the physical activity in the past 7 days, and Sedentary Behavior Record assessing the daily patterns of activities exhibited in a sitting posture. To match the measurement phase between the device-based (Actigraph wGT3X-BT®) and self-reported assessments of physical activity and sedentary behavior, the Global physical Activity Questionnaire will be completed on the day that participants remove the Actigraph wGT3X-BT®, and the Sedentary Behavior Record will be completed on four consecutive days (two week and two weekend days) of participants' choice during the 7 days device wearing. -These questionnaires will be administered electronically after the baseline physical assessment, however, if the participant prefers a paper copy this option will be available at the baseline evaluation meeting. Consented participants who have completed baseline assessments will then be randomized.

Group 1: Tai Chi Intervention group (20 total participants) This group will be instructed to follow a Tai Chi program led by a certified teacher starting 8 weeks prior to their scheduled surgery date. To facilitate physical distancing in accordance to the current COVID-19 restrictions and while optimizing the quality of the intervention, the Tai Chi program will be administered virtually (via Zoom) by combining both supervised and unsupervised session. The program will be organized via a twofold approach: 1) a 60-minute supervised practice will be administered 2 days per week to patient participants and caregivers, if applicable. This session will be offered live via password protected Zoom and will be led by a Tai Chi instructor certified in WaQi teaching. It will include a warmup, agility training, meditation, slow movement, and meditation for cooling down; and 2) a 15-minute home-based program will be administered via an un-supervised online teaching module five days/week. It involves meditation, slow movement, and agility training and will be delivered via a webpage with a subscription for each patient participant and caregiver, if applicable.

Group 2: Usual activity group (20 total participants) This group will be instructed to maintain their physical activity levels for a total of 8 weeks. They will be provided with printed materials from Prostate Cancer Canada about prostate cancer management. They will receive an 8-week online Tai Chi teaching module subscription at the end of the study.

Participants in both control and intervention arms will wear the Actigraph wGT3X-BT® accelerometer for one week and complete two questionnaires (Global Physical Activity Questionnaire, and Sedentary Behavior Record) at 6 weeks after baseline (2 weeks prior to surgery). Participants will repeat five questionnaires (Pittsburgh Sleep Quality Inventory, SF-36, Hospital Anxiety and Depression Scales, Brief Pain Inventory, the urinary and sexual domains of the Expanded Prostate Cancer Index Composite-50 [spousal version for spousal caregivers]) and physical function tests at the 6 weeks after baseline (2 weeks prior to surgery), 6 weeks post-surgery (follow-up visit to review pathology and check PSA) and 12 weeks (or 3 months) post-surgery (PCC follow-up visit). Participants will complete additional Hospital Anxiety and Depression Scales at surgery day and at 2 weeks post-surgery (follow-up visit for catheter removal). Finally, frailty will be derived through a modified frailty index using data extracted from electronic medical charts at 12 weeks (or 3 months).

At the completion of the intervention/study 25 qualitative interviews will be conducted to assess the barriers and facilitators related to implementing the online Tai Chi intervention targeting five domains of the Consolidated Framework for Implementation Research (CFIR): intervention characteristics, outer setting, inner setting, characteristics of the individuals involved, and the process of implementation. Multiple stakeholders including 10 patient participants, 10 caregiver participants, the Tai Chi instructor and five healthcare providers will be interviewed to evaluate CFIR domains that are relevant to them. The interview will be semi-structured in design and will last approximately 1-hour via password-protected Zoom and recorded.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

* Must speak English.
* Scheduled and awaiting radical prostatectomy for prostate cancer
* Not previously treated for prostate cancer, including radiation therapy to the pelvis, major pelvic surgery, or placement of a penile implant or artificial urinary sphincter
* No known urethral stricture or colostomy or chronic urinary catheterization
* No medical or current psychiatric disorders that precludes their participation in the
* Permission to exercise from their primary physicians
* Not currently practicing Tai Chi or related activities that involve mindfulness practice
* Has access to a computer or tablet, reliable internet and the skills/knowledge to use email, complete online questionnaire and attend Zoom meetings.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Participant recruitment rate | 8 weeks
  Evaluate the percentage of patients willing to participate in the intervention among eligible patients approached
Intervention uptake ratio | 8 weeks
  A ratio of the number of participants who actively participated in the intervention against the total number of participants in the intervention group will be assessed.
Adherence to intervention | 8 weeks
  Calculate percentage of intervention completions based on the numbers of attended sessions and the duration of attendance
Reasons for withdrawal | 8 weeks
  Will record reasons for withdrawal for those participants that withdraw from the study, when applicable.
Adverse events | 8 weeks
  Will record all adverse events that occur over the course of the intervention, if applicable.
Intervention barriers and facilitators | 8 weeks
  Qualitative data collection and interview guide development will follow the CFIR methodology to assess the intervention barriers and facilitators under five domains: intervention characteristics (key attributes of interventions), outer setting (factors outside the implementation organization), inner setting (factors within the implementation organization), characteristics of the individuals involved (perceptions, attitudes, and motivation of individuals), and the process (strategies to support implementation)

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Inventory (PSQI) | 5 months
  Measure of sleep quality captured by a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Nineteen individual items (scored on scale from 0-3) generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score (range: 0-21) where a higher score corresponds to lower sleep quality.
Short Form-36 (SF-36) | 5 months
  Measure quality of life assessed SF-36 measures eight scales including 36 items on: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH); Overall score between 0-100, where lower scores correspond to greater disability.
General Anxiety Disorder 7-item Scale (GAD-7) | 5 months
  7-item anxiety scale where responders are asked to rate the frequency of anxiety symptoms in the last 2 weeks on a Likert scale ranging from 0-3. Items are summed to provide a total score ranging from 0-21, where a higher score corresponds to greater anxiety.
Patient Health Questionnaire (PHQ-9) | 5 months
  the PHQ-9 is the depression module of the Patient Health Questionnaire (PHQ), which is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 module scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day) for a total score ranging from 0-27, where higher scores correspond to greater levels of depression.
Brief Pain Inventory (BPI) | 5 months
  Measure of pain he BPI is an 11-item questionnaire that consists of four 0-to-10 numeric rating scale (NRS) items asking patients to rate their pain at its "worst in the last 24-hours," "least in the last 24-hours," "average," and "now," with a 0 indicating "no pain" and 10 representing "pain as bad as you could imagine." The remaining seven BPI items probe the degree to which pain interferes with general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life, again using a 0-to-10 NRS. For these interference items, 0 represents "does not interfere" and 10 indicates "interferes completely." The arithmetic mean of the 4 pain severity items is taken as a measure of pain severity, and the seven interference items can be used as a measure of pain interference (higher score = higher pain severity/pain interference)
Expanded Prostate Cancer Index Composite (EPIC) | 5 months
  Expanded Prostate Cancer Index Composite for Clinical Practice is a 1-page, 16-item questionnaire that we constructed to measure urinary incontinence, urinary irritation, and the bowel, sexual and hormonal health related quality of life domains. Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale with higher scores representing better Health-Related Quality of Life (HRQOL).
Physical function | 5 months
  Physical function will be assessed through handgrip strength measured by a dynamometer, six minute walk test measured with a stopwatch and measuring tape, and four functional tests in accordance with the US CDC STEADI (Stopping Elderly Accidents, Deaths & Injuries) older adults fall prevention program that consists of 30-seconds chair stand test, 4-stage balance test, timed up and go test, and orthostatic blood pressure. These measures are standardized and validated gait, strength and balance assessment and predictors of physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yang, PhD, Principal Investigator — Alberta Health services
Locations (1):
- Prostate Cancer Centre, Calgary, Alberta, Canada